CLINICAL TRIAL: NCT03171974
Title: Ultrasound Guided Treatment of Steroids for Capsular Contracture in Patients With Reconstructed/Augmented Breast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Muhamad Mansur, Principal investigator, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0213-17-RMC
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Capsular Contracture, Implant
Keywords: breast capsular contructure
MeSH Terms: conditions — Implant Capsular Contracture | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: one treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): The treatment group will be injected with dexamethasone instracapsular under US according to our built protocol.
  Interventions: Drug: Dexamethasone; Device: US

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone will be injected intracapsular under US
Device: US — dexamethasone will be injected intracapsular under US

SUMMARY:
Ultrasound guided treatment of steroids for capsular contracture in patients with reconstructed/augmented breast

DETAILED DESCRIPTION:
The aim of this study is to evaluate ultrasound (US)-guided treatment of capsular contracture (CC) in patients with reconstructed/ augmented breast.

Capsular contraction is the one of the most common complications of both esthetic and reconstructive breast surgery with an incidence of 0.5-30% and 1-38%, respectively. In irradiated patients the incidence is higher, in the range of 30-67%. It appears most commonly in the first year but in some patients, belated capsular contracture has been noticed. The more severe forms of contraction, Baker grades 3 and 4 with a firm often deformed and painful breast, have been shown to recur as often as 67% after capsulotomy

steroid injection has been demonstrated to be effective for the treatment of this condition.

20-30 female with grade III\IV CC will be included. Patients will be treated with peri-implant US-guided injection of Dexamethasone

The purpose of our study is to use a longer acting steroid (Dexamethasone) injected intra capsular with US-guide. By that getting a better effect on the level of fibrosis.

This Clinical study will be conducted in the tertiary academic Rabin Medical Center.

Several measures will be taken, including: capsular contracture grading by two plastic surgeons, a VAS-score of breast pain, maximal capsular thickness (MCT) in sonography

ELIGIBILITY:
Inclusion Criteria:

• female patient with grade 3-4 capsular contraction after alloplastic breast reconstruction\ augmentation

Exclusion Criteria:

* intake of steroids, anti-inflammatory, anti-coagulate or immunomodulatory medications on a regular basis
* Patients with skin atrophy of the breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
reducing maximum capsular thickness (MCT) | 3.5 years
  measured by ultrasound
reduce pain | 3.5 years
  pain assessed with visual analogue score (pain-VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Mansour, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, IL, Israel

IPD SHARING:
Plan to Share IPD: Yes